CLINICAL TRIAL: NCT04323306
Title: A Two-part, Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetic Profile of Ascending Single Doses of MMV533, Including a Pilot Food Evaluation in Healthy Participants.
Brief Title: A Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetic Profile of a Single Doses of MMV533.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Nucleus Network Ltd (Other); Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV-MMV533_19_01
Record Dates: First submitted 2020-03-12; First posted 2020-03-26 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Malaria
Keywords: Safety; Tolerability
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Part 1: 8 participants per cohort for 7-8 cohorts (56-64 participants total). Single ascending dose commencing at 5 mg with maximum 400 mg as determined by Safety Review Committee (SRC).
  Part 2:
  Open label, 2-period cross-over, randomized, pilot food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV533
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple for part 1. Double-blind, randomized, placebo-controlled, sequential ascending single dose study Open label for part 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 SAD (Active Comparator): 5 mg MMV533 with single ascending dose
  Interventions: Drug: MMV688533
- Cohort 2 SAD (Active Comparator): Single ascending dose to be determined after SRC review of previous cohort.
  Interventions: Drug: MMV688533
- Cohort 3 SAD (Active Comparator): Single ascending dose to be determined after SRC review of previous cohort.
  Interventions: Drug: MMV688533
- Cohort 4 SAD (Active Comparator): Single ascending dose to be determined after SRC review of previous cohort.
  Interventions: Drug: MMV688533
- Cohort 5 SAD (Active Comparator): Single ascending dose to be determined after SRC review of previous cohort.
  Interventions: Drug: MMV688533
- Cohort 6 SAD (Active Comparator): Single ascending dose to be determined after SRC review of previous cohort.
  Interventions: Drug: MMV688533
- Cohort 7 SAD (Active Comparator): Single ascending dose to be determined determine after SRT review of previous cohort. Dose will not exceed 400 mg.
  Interventions: Drug: MMV688533
- Part 2: Food Effect (Active Comparator): Open label, 2-period cross-over, randomized, pilot food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV533 determined to be safe in Part 1.
  Interventions: Drug: MMV688533

INTERVENTIONS:
Drug: MMV688533 — Investigational medicinal product

SUMMARY:
Phase 1, single -centre study in 2 parts. The study designs for each part are well established for first-in-human studies and are appropriate to assess safety, tolerability and preliminary pharmacokinetics.

DETAILED DESCRIPTION:
Part 1:

Double-blind, randomized, placebo-controlled, sequential ascending single dose study in healthy adult participants, 7 cohorts, and 1 additional cohort may be considered if needed according to the observed safety, tolerability, and pharmacokinetics results.

A sentinel dosing strategy will be implemented at each dose level to ensure the best conditions of safety. Each cohort will be divided into at least 2 subgroups. The first group (sentinel cohort) will include 2 participants that will be dosed on the first day, with 1 participant receiving MMV533 and 1 participant receiving placebo. The safety and tolerability data from the sentinel cohort up to and including 96 hours post-dose will be reviewed by the Principal Investigator, the Medical Monitor and the Sponsor´s Medical Director. Following a satisfactory safety review, dosing of the remaining participants in the cohort may proceed.

Part 2:

Open label, 2-period cross-over, randomized, pilot food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV533 to healthy male and female participants aged between 18-55 years old. Part 2 may be conducted in parallel to or after completion of Part 1 at the discretion of the SRC. The dose will be selected by the SRC based on PK and safety results obtained in Part 1 and also taking into account the human efficacious dose/exposure predicted from preclinical efficacy studies in rodent malaria models.

ELIGIBILITY:
Inclusion Criteria

1. Males and females (of childbearing and non-childbearing potential) , between 18 and 55 years of age, inclusive. Women of childbearing potential (WOCBP) must use highly effective methods of birth control (see Inclusion #3).
2. Females of non-childbearing potential:

   1. Natural (spontaneous) post-menopausal defined as being amenorrhoeic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level (FSH) >25 IU/L (or at the local laboratory levels for post-menopause)
   2. Premenopausal with irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy or salpingectomy at least 6 months before screening (as determined by participant medical history)
3. Women of childbearing potential that have or may have male sexual partners during the course of the study must agree to the use of a double method of contraception of a highly effective method of birth control combined with a barrier contraceptive (condom) when appropriate from screening visit to until 60 days after the last dose of IMP (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose of IMP. This duration is based on the predicted half-life of IMP, and may be amended once the actual half-life is calculated during this study). Note: Highly effective birth control methods include: combined (oestrogen and progestogen containing) oral/intravaginal/transdermal hormonal contraception associated with inhibition of ovulation, progestogen-only oral/injectable/implantable hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, or sexual abstinence or same sex relationship.
4. Male participants who have, or may have female sexual partners during the course of the study must agree to use a double method of contraception including condom plus diaphragm, or condom plus stable insertable (implant or IUD), injectable, transdermal or combination oral contraceptive by the female partner, from the time of informed consent through to 90 days after the last dose of the IMP (covering a full spermatogenesis cycle of 60 days starting after 5 half-lives of last dose of IMP. This duration is based on the predicted half-life of IMP, and may be amended once the actual half-life is calculated during this study).

   Abstinent male participants must agree to start a double method if they begin a sexual relationship with a female during the trial, and through to 90 days after the last dose of the IMP. Male participants with female partners that are surgically sterile or post-menopausal (defined as being amenorrhoeic for at least 12 months without an alternative medical cause), or male participants who have undergone sterilisation and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above described methods of contraception. Male participants must also agree not to donate sperm up to 3 months after dosing with the IMP.
5. Total body weight greater than or equal to 50 kg, and body mass index (BMI) between 18 and 32 kg/m2 inclusive.
6. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
7. Normal vital signs after 5 minutes resting in supine position:

   * Systolic blood pressure (SBP) - 90-140 mmHg,
   * Diastolic blood pressure (DBP) - 40-90 mmHg,
   * Heart rate (HR) 40-100 bpm.
8. Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges for both males and females: QT ≤ 500 msec, QTcF ≤450 msec, QTcB ≤450 msec, and PR interval ≤210 msec; and normal ECG tracing unless the Principal Investigator or delegate considers an ECG tracing abnormality to be not clinically significant.
9. Having given written informed consent prior to undertaking any study-related procedure.
10. Available for the duration of the study and for 2 weeks following the End of Study visit.
11. In the opinion of the Principal Investigator or delegate, the individual has a high probability of adherence with and completion of the study, and willing and able to withdraw and refrain from restricted medications.
12. Fluent in English and able to understand and comply with written and verbal protocol-related requirements.
13. Willing to defer blood donations to a blood service for a minimum of 6 months after the End of Study visit.

Exclusion Criteria

1. Haematology, biochemistry or urinalysis results that are abnormal/outside of laboratory normal reference ranges AND are either:

   * considered clinically significant by the Principal Investigator or delegate; OR
   * considered not clinically significant by the Principal Investigator or delegate BUT ARE ALSO outside of the Sponsor-approved clinically acceptable laboratory ranges in Appendix 1 of the protocol.

   NOTE: Participants are not excluded if abnormal/out of laboratory normal reference range results are considered not clinically significant by the Principal Investigator or delegate AND are within the ranges specified in Appendix 1 of the protocol of .
2. Positive serum pregnancy test at screening, positive urine pregnancy test upon admission or at other timepoints as specified by schedule of assessments.
3. Male participants with a female partner(s) who is (are) pregnant or lactating from the time of the administration of study medication.
4. Any history or presence of clinically relevant cardiovascular, broncho-pulmonary, gastrointestinal, hepatic/ gallbladder*/ bile duct, renal, metabolic, haematological, neurological, musculoskeletal/rheumatologic, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness. *including medical history of asymptomatic gallbladder stones.
5. Any gastrointestinal surgery or any condition or disease that could affect drug absorption, distribution or excretion (eg, gastrectomy, cholecystectomy, diarrhoea).
6. Severe recurring headaches (cluster or migrainous headaches) requiring prescription medication/s. History of recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
7. Participation in any research study involving blood sampling (more than 450 mL/unit of blood) or blood donation during the 8 weeks prior to IMP administration (Parts 1 and 2).
8. Any documented evidence of current or past cardiovascular disease including cardiac arrhythmias or family history of congenital long QT syndrome, Brugada syndrome, or unexplained sudden cardiac death. Symptomatic postural hypotension at screening (confirmed on two consecutive readings), irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 min when changing from supine to standing position.
9. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies, or any history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing. Participants with seasonal allergies/hay fever or allergy to animals or house dust mite that are untreated and asymptomatic at the time of dosing can be enrolled in the trial.
10. History of convulsion (including drug or vaccine-induced episodes). A medical history of a single febrile convulsion during childhood is not an exclusion criterion.
11. History of substance use disorder(s) within 5 years of screening, including alcohol consumption of more than 40g/4 units/4 standard drinks per day or any prior intravenous use of an illicit substance.
12. Smoked >1 pack of cigarettes per day for >10 years, or who currently (within 14 days prior to IMP administration (Parts 1 and 2) smokes >5 cigarettes per day.
13. Any medication (including herbal such as St John´s Wort, vitamin supplements and over the counter [OTC]) within 5 half-lives prior to IMP administration (Parts 1 and 2), except occasional intakes (for acute pain) of ibuprofen at doses up to 1.8g/day, paracetamol at doses up to 4g/day, acetylsalicylic acid (300 to 650 mg orally every 4 to 6 hours as needed Maximum dose: 4g in 24 hours), diclofenac (diclofenac potassium liquid-filled capsules: 25mg orally 4 times a day; diclofenac free acid capsules: 18 or 35 mg orally 3 times a day; diclofenac potassium immediate-release tablets: 50mg orally 3 times a day [initial dose of 100mg orally followed by 50mg oral doses acceptable if required for better relief]) and contraceptives.
14. Any individual who, in the judgement of the Principal Investigator or delegate, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
15. Any individual in the exclusion period of a previous study according to applicable regulations.
16. Any individual who cannot be contacted in case of emergency.
17. Any individual who is the Investigator, or delegates, research assistant, pharmacist, study coordinator, project manager, or other staff thereof, directly involved in conducting the study.
18. Any individual without a good peripheral venous access.
19. Participation in any investigational product study within the 12 weeks preceding IMP administration (Parts 1 and 2) or 5 times the half-life of the Investigational product, whichever is longer.
20. Positive serology test for hepatitis B (positive HB sAG or anti-HBc Ab), hepatitis C (anti-HCV) or human immune deficiency virus (HIV) (positive for anti-HIV1 and anti-HIV2 Ab).
21. Positive urine drug test at screening or prior to IMP dosing. Any drug from the list of drugs tested unless there is an acceptable explanation to the Principal Investigator or delegate (eg, participant has stated in advance that they consumed a prescription of over the counter product which contained the detected drug) and/or the participant has a negative urine drug screen on retest. Any participant tested positive for paracetamol at screening may still be eligible for study participation, at the Principal Investigator's or delegate's discretion.
22. Positive alcohol screen at screening or prior to IMP dosing.
23. Any consumption of citrus fruits (grapefruit, Seville oranges) or their juices within 5 days prior to IMP administration.
24. Use of antidepressant medication in the past 12 months prior to IMP administration in Part 1 and 2.
25. Individuals with history of schizophrenia, bipolar disorder psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis including generalised anxiety and obsessivecompulsive disorders.
26. Individuals who have been hospitalised within five years prior to enrolment for either a psychiatric illness or due to danger to self or others.
27. History of an episode of mild/moderate depression lasting more than 6 months that required pharmacological therapy and/or psychotherapy within the last 5 years; or any episode of major depression. The Beck Depression Inventory (BDIII) will be used as a validated tool for the assessment of depression at screening. In addition to the conditions listed above, individuals with a score of 20 or more on the BDI-II and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. These individuals will be referred to a general practitioner or medical specialist as appropriate. Individuals with a BDI-II score of 17 to 19 may be enrolled at the discretion of an Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the individual or to the execution of the trial and interpretation of the data gathered.
28. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer considered treated and cured), treated or untreated, within 5 years of screening, regardless of whether there is no evidence of local recurrence or metastases.
29. Any vaccination within 28 days of screening.
30. Any medical condition that in the opinion of the Principal Investigator or delegate would jeopardize the individual's involvement in the study.

    Specific to Part 2 only:
31. Any individual who, in the opinion of the Principal Investigator or delegate, would be unwilling or unable to consume the pre-dose test meal during the fed arm.
32. Individuals with food intolerance or food allergy are excluded. Vegetarian individuals must be excluded, unless they agree to eat a full diet during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network Corporate
Locations (1):
- Nucleus Network Corporate, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bestgen B, Jones S, Thathy V, Kuemmerle A, Barcelo C, Haouala A, Gossen D, Marx MW, Di Resta I, Szramowska M, Webster RA, Llewellyn S, Ritacco DA, Yeo T, Leroy D, Barber BE, Fidock DA, Griffin P, Lickliter J, Chalon S. Safety, tolerability, pharmacokinetics, and antimalarial activity of MMV533: a phase 1a first-in-human, randomised, ascending dose and food effect study, and a phase 1b Plasmodium falciparum volunteer infection study. Lancet Infect Dis. 2025 May;25(5):507-518. doi: 10.1016/S1473-3099(24)00664-9. Epub 2024 Dec 18. PMID 39708824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A: Up to 64 participants planned, 7 ascending single doses of MMV533 were planned, with up to 1 additional dose level if required. Starting dose 5 mg.
  Part B: 8 participants planned.
  The study incorporated the use of an adaptive design to allow for flexibility in the conduct of the study
Groups:
- Cohort 1 SAD: 5 mg MMV533
  MMV688533: Investigational medicinal product
- Cohort 2 SAD: 10 mg MMV533
  MMV688533: Investigational medicinal product
- Cohort 3 SAD: 20 mg MMV533
  MMV688533: Investigational medicinal product
- Cohort 4 SAD: 50 mg MMV533
  MMV688533: Investigational medicinal product
- Cohort 5 SAD: 100 mg MMV533
  MMV688533: Investigational medicinal product
- Cohort 6 SAD: 160 mg MMV533
  MMV688533: Investigational medicinal product
- SAD Placebos: Pooled placebos
- Part 2: Food Effect; MMV 533 (30mg) Fasted/Fed: 4 participants were randomised and received MMV 533 (30mg) in Fasted state before cross-over to be administered 30 mg of IMP Fed state, 28 days post initial dose
- Part 2: Food Effect; MMV 533 (30mg) Fed/Fasted: 4 participants were randomised and received MMV 533 (30mg) in Fed state before cross-over to be administered 30 mg of IMP Fasted state, 28 days post initial dose
Period: Overall Study
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | SAD Placebos | Part 2: Food Effect; MMV 533 (30mg) Fasted/Fed | Part 2: Food Effect; MMV 533 (30mg) Fed/Fasted
Started | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 4 | 5
Completed | 5 | 6 | 6 | 6 | 6 | 7 | 9 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1-MMV533 5 mg: 6 participants were randomised and received 5 mg administered in fasting condition
- Cohort 2 MMV533 10 mg: 6 participants were randomised and receive 10 mg in fasting condition
- Cohort 3 MMV533 20 mg: 6 eligible participants were randomised and received 20 mg in fasting condition
- Cohort 4 MMV533 50 mg: 6 eligible participants were randomised and received 50 mg in fasting condition
- Cohort 5 MMV533 100 mg: 6 eligible participants were randomised and received 100 mg in fasting condition
- Cohort 6 MMV533 160 mg: 6 eligible participants were randomised and received 160 mg in fasting condition
- Placebo: 12 participants across 6 cohorts were randomised and received placebo administered in fasting condition
- Total: Total of all reporting groups
Arm/Group | Cohort 1-MMV533 5 mg | Cohort 2 MMV533 10 mg | Cohort 3 MMV533 20 mg | Cohort 4 MMV533 50 mg | Cohort 5 MMV533 100 mg | Cohort 6 MMV533 160 mg | Placebo | Part 2: Food Effect; MMV 533 (30mg) Fasted/Fed | Part 2: Food Effect; MMV 533 (30mg) Fed/Fasted | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 4 | 5 | 59
Age, Continuous [Median (Standard Deviation); unit: years] | 26.0 (3.34) | 34.0 (6.18) | 21.5 (5.57) | 30.0 (8.14) | 23.0 (11.69) | 37.0 (7.69) | 25.5 (8.51) | 32.0 (7.41) | 28.0 (7.33) | 28.0 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 3 | 1 | 3 | 6 | 2 | 2 | 27
  Male | 2 | 2 | 4 | 3 | 5 | 5 | 6 | 2 | 3 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 6 | 3 | 6 | 5 | 6 | 7 | 12 | 4 | 5 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 3 | 3 | 1 | 5 | 0 | 2 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 5 | 5 | 5 | 3 | 3 | 5 | 7 | 3 | 3 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index [Median (Standard Deviation); unit: kg/m2] | 22.50 (2.176) | 24.95 (3.144) | 23.00 (1.218) | 25.80 (2.769) | 23.95 (2.737) | 23.15 (3.261) | 23.50 (1.969) | 24.00 (2.598) | 25.90 (1.503) | 23.90 (2.413)

OUTCOME MEASURES:

1. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Assessment of adverse events (AEs) /treatment-emergent adverse events (TEAEs) (treatment phase for Part 1 and 2 defined as from IMP administration up to and including EOS).
Time Frame: Safety data will be evaluated from baseline until 28 days after IMP/placebo administration
Population: Part 1: Up to 64 participants planned, 53 randomised with 50 administered IMP. All 53 analysed in Full Analysis Set (FAS), 50 (dosed) analysed in Safety Set and 38 (administered MMV533) analysed in the PK set.
  Part 2: 8 planned, 9 randomised and received at least one dose; 9 analysed in Safety Set. 6 participants in the PK completer subset (both periods completed, no major PDs) and 9 participants in the PK analysis subset (at least one period completed with no major PDs).
Measure: Number; unit: participants
Groups:
- Cohort 1 SAD: 5 mg MMV533
  6 participants were randomized to receive MMV533
- Cohort 2 SAD: 10 mg MMV533
  6 participants were randomized to receive MMV533
- Cohort 3 SAD: 20 mg MMV533
  6 participants were randomized to receive MMV533
- Cohort 4 SAD: 50 mg MMV533
  6 participants were randomized to receive MMV533
- Cohort 5 SAD: 100 mg MMV533
- Cohort 6 SAD: 160 mg MMV533
  8 participants were randomized to receive MMV533
- Placebo: Placebo across Cohorts 1-6
- Part 2: Food Effect: MMV533 30mg Fasted
- Part 2 - Food Effect: MMV533 30mg Fed
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect | Part 2 - Food Effect
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
participants
  Participants with at least one TEAE | 5 | 3 | 7 | 4 | 3 | 4 | 6 | 5 | 6
  Participants with at least one IMP-related TEAE | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
  Participants with at least one Procedure-related TEAE | 2 | 0 | 1 | 2 | 2 | 0 | 1 | 4 | 0

2. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Haematology: change from baseline
Time Frame: Change from baseline to 28 days post dose in Part 1 of the study and 21 days post dose in Part 2, Food effect study
Population: For Part A overall, 50 (94.3%) participants were included in the Safety Set whereas for Part B, all 9 (100%) participants were included, and no participants were excluded from the Safety Set.
Measure: Mean (Standard Deviation); unit: 10^9 *cells*/L
Groups:
- Cohort 5 SAD: 100 mg MMV533
  6 participants were randomized to receive MMV533
- Part 2: Food Effect: Period 1: 8 participants fasted and administered 30 mg of IMP
- Part 2: Food Effect Cohort: Period 2: 9 participants fed and administered 30 mg of IMP
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect | Part 2: Food Effect Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
10^9 *cells*/L
  Basophils | -0.02 (0.04) | 0.03 (0.05) | 0.00 (0.00) | 0.00 (0.00) | 0.03 (0.05) | 0.00 (0.06) | 0.01 (0.05) | -0.01 (0.04) | 0.00 (0.05)
  Eosinophils | 0.02 (0.08) | -0.03 (0.08) | 0.00 (0.11) | -0.02 (0.08) | -0.02 (0.08) | -0.01 (0.07) | -0.04 (0.09) | -0.04 (0.09) | -0.03 (0.05)
  Lymphocytes | -0.40 (0.24) | -0.18 (0.26) | -0.28 (0.15) | -0.35 (0.36) | -0.33 (0.26) | -0.24 (0.59) | -0.18 (0.35) | -0.10 (0.21) | -3.4 (0.59)
  Monocytes | 0.02 (0.17) | -0.03 (0.05) | 0.08 (0.08) | -0.02 (0.08) | -0.08 (0.08) | -0.01 (0.12) | 0.04 (0.09) | 0.04 (0.05) | -0.01 (0.10)
  Neutrophils | 0.12 (1.96) | -0.25 (0.72) | 0.33 (0.53) | 0.47 (0.90) | -0.97 (2.29) | 0.23 (0.44) | 0.09 (1.88) | 0.14 (0.75) | -0.10 (0.92)
  Platelets | 20.0 (25.3) | 24.0 (20.6) | 5.0 (21.8) | 2.5 (13.6) | 4.8 (36.7) | 18.4 (26.0) | 8.9 (26.6) | -3.3 (6.2) | 28.3 (12.6)
  Leukocytes | -0.20 (2.04) | -0.52 (0.87) | 0.10 (0.49) | 0.07 (1.13) | -1.33 (2.35) | 0.00 (0.95) | -0.12 (2.07) | 0.03 (0.90) | -0.48 (0.96)

3. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Biochemistry: number of participants with elevated Total Bile Acids considered as Clinically significant abnormalities
Time Frame: 24 hours to 648 hours post dose
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Food Effect_Fasted: Period 1: 8 Participants Fasted and given 30 mg of IMP
- Part 2: Food Effect cohort_Fed: Period 2: 9 Participants Fed and given 30 mg of IMP
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
Participants
  24 hour 24 hour | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
  72 hour | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
  168 hour | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  312 hour | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  480 hour | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  648 hour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Urinalysis: parameters assessed: bilirubin, glucose, ketones, leucocytes, nitrite, blood, protein, urobilinogen, pH.
  Number of participants with clinically significant findings.
Time Frame: Part 1: 28 days post IMP administration and for Part 2: 21 days post IMP administration
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Vital signs: respiratory rate supine and standing. Change from baseline.
Time Frame: Part 1 is 28 days post IMP and for Part 2, 21 days post IMP administration
Measure: Median (Standard Deviation); unit: Change in the number of breaths/minute
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
Change in the number of breaths/minute
  Respiratory Rate (Supine) (breaths/min) | 0.0 (1.6) | 0.0 (2.2) | 0.0 (1.5) | 2.0 (4.1) | 2.0 (1.5) | 2.0 (2.5) | 0.0 (3.2) | 0.0 (1.8) | 0.0 (1.7)
  Respiratory Rate (Standing) (breaths/min) | 0.0 (1.5) | 0.0 (4.1) | 0.0 (1.8) | 2.0 (2.8) | 1.0 (2.0) | 2.0 (2.9) | 0.0 (3.4) | 2.0 (2.3) | 2.0 (1.0)

6. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Vital signs: heart rate supine and standing. Change from baseline.
Time Frame: Part 1 is 28 days post IMP and for Part 2, 21 days post IMP administration
Measure: Median (Standard Deviation); unit: Change in the number of beats/minute
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
Change in the number of beats/minute
  Heart Rate (beats/min)- Supine | 0.5 (8.5) | -5.0 (7.5) | 9 (8.7) | 4 (12.6) | 6 (11.1) | 0.9 (11.1) | -1 (7.2) | 6.5 (8.3) | 4 (11.3)
  Heart Rate (beats/min)- Standing | 22 (13) | 8 (9.4) | 25 (13.5) | 16.5 (10.5) | 17.5 (10.3) | 16 (11.8) | 11.9 (19.5) | 14 (6) | 12.5 (13.1)

7. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Measurements of 12-lead triplicate ECG: QTcB and QTcF interval prolongations.
Time Frame: Part 1: 28 days post IMP whereas for Part 2: 21 days post IMP administration
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
Participants
  QTcB Interval, Aggregate (ms) Prolongation >30 ms | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval, Aggregate (ms)Prolongation >60 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  QTcB Interval, Aggregate (ms) >450 ms | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, Aggregate (ms) Prolongation >30 ms | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, Aggregate (ms)Prolongation >60 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, Aggregate (ms) >450 ms | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Biochemistry: number of participants with Low Hemoglobin considered as Clinically significant abnormality
Time Frame: 24 hours to 648 hours post dose
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 12 | 8 | 9
Participants
  24 hour 24 hour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  72 hour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  168 hour | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 2 | 0
  312 hour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  480 hour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  648 hour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Vital signs: blood pressures, supine and standing. Change from baseline.
Time Frame: Part 1 is 28 days post IMP and for Part 2, 21 days post IMP administration
Measure: Median (Standard Deviation); unit: mm Hg
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 9
mm Hg
  Systolic Blood Pressure (mmHg)-Supine | 3 (8.6) | 22.5 (7.5) | 3 (13.9) | 4 (6.1) | 2 (9.3) | 5 (10.6) | 3 (8.5) | -0.5 (7.3) | -2.5 (10.7)
  Systolic Blood Pressure (mmHg)-Standing | 4 (17) | 11 (10.6) | -0.5 (10.7) | 4.5 (4.8) | -4.5 (11.8) | 2 (13.3) | 1 (10) | 0.5 (5.9) | 4 (9.6)
  Diastolic Blood Pressure (mmHg)- Supine | -3.5 (6) | 2 (7) | 0 (8.5) | 0.5 (4.7) | -2 (7) | 2 (5.) | 0 (7.1) | -2 (6.1) | -1.5 (8.1)
  Diastolic Blood Pressure (mmHg)- Standing | 9.5 (5) | 9 (7.3) | 7.5 (7) | -1 (5.2) | 5 (6.2) | 11.8 (9.3) | 5 (6.1) | 7.5 (7.4) | 7 (2.1)

10. Primary Outcome: The Tolerability and Safety of Ascending Single Oral Doses of MMV533
Description: Vital signs: body temperature. Change from baseline.
Time Frame: Part 1 is 28 days post IMP and for Part 2, 21 days post IMP administration
Measure: Median (Standard Deviation); unit: Celsius degree
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Placebo | Part 2: Food Effect_Fasted | Part 2: Food Effect cohort_Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 9
Celsius degree | 0.25 (0.56) | 0.5 (0.81) | 0.05 (0.36) | 0.35 (0.66) | -0.1 (0.61) | -0.10 (0.39) | -0.1 (0.51) | -0.1 (0.7) | 0 (0.4)

ADVERSE EVENTS:
Time Frame: AEs were collected until EOS i.e. up to Day 28 in Part A and up to Day 42 in Part B.
Description: AEs include Serious Adverse Events (SAE) and Adverse Events for Special Interest (AESI).
  Results from placebo are pooled together because there were no events recorded for any of the participants receiving the placebo.
Groups:
- Cohort 2 SAD: 10 mg
  MMV688533: Investigational medicinal product
- Cohort 3 SAD: 20 mg
  MMV688533: Investigational medicinal product
- Cohort 4 SAD: 50 mg
  MMV688533: Investigational medicinal product
- Cohort 5 SAD: 100 mg
  MMV688533: Investigational medicinal product
- Cohort 6 SAD: 160 mg
  MMV688533: Investigational medicinal product
- Part A Placebo Participants: All placebo pooled together
- Part B Fasted: 30 mg
  Open label, 2-period cross-over, randomized, pilot food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV533 determined to be safe in Part 1.
  MMV688533: Investigational medicinal product
- Part B Fed: 0 mg
  Open label, 2-period cross-over, randomized, pilot food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV533 determined to be safe in Part 1.
  MMV688533: Investigational medicinal product
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Cohort 3 SAD | Cohort 4 SAD | Cohort 5 SAD | Cohort 6 SAD | Part A Placebo Participants | Part B Fasted | Part B Fed
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/12 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/8 | 0/12 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/12 | 0/8 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 SAD (N=6) | Cohort 2 SAD (N=6) | Cohort 3 SAD (N=6) | Cohort 4 SAD (N=6) | Cohort 5 SAD (N=6) | Cohort 6 SAD (N=8) | Part A Placebo Participants (N=12) | Part B Fasted (N=8) | Part B Fed (N=9)
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
No limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT04323306/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04323306/SAP_001.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT04323306/ICF_002.pdf